CLINICAL TRIAL: NCT01754363
Title: Short, Medium and Long Term Survivorship of Attune Primary Knee Prosthesis
Brief Title: Survivorship of Attune Primary Total Knee Prosthesis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10008
Record Dates: First submitted 2012-12-18; First posted 2012-12-21 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Noninflammatory Degenerative Joint Disease
Keywords: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Attune Primary Total Knee Replacement (Experimental): Subjects will receive one of the following Attune total knee implants:
  Cruciate retaining fixed bearing (CR FB) Cruciate retaining rotating platform (CR RP) Posterior stabilized fixed bearing (PS FB) Posterior stabilized rotating platform (PS RP)
  Interventions: Device: Attune Primary Total Knee Replacement

INTERVENTIONS:
Device: Attune Primary Total Knee Replacement — Patients will undergo a primary total knee replacement using one of the four configurations of the Attune knee (CR FB, CR RP, PS FB, PS RP).

SUMMARY:
This post-marketing investigation will evaluate the long term (up to 15 years) survivorship of the Attune Primary Knee Prosthesis in patients with non-inflammatory degenerative joint disease. Data from Subjects who receive one of four knee configurations will be pooled to establish a contemporary dataset.

DETAILED DESCRIPTION:
Approximately 30 sites, worldwide, will recruit 1200 patients (1200 knees). Each study site is expected to enroll approximately 50 patients (50 knees). An additional 10 subjects per site may be recruited at sites which have Sub-Investigators participating in the study. Cohort reallocation is permitted. There is no control group. One thousand two hundred (1200) Subjects will be stratified into 4 subgroups of 300: cruciate retaining fixed bearing(CR FB), cruciate retaining rotating platform (CR RP), posterior stabilized fixed bearing (PS FB), and posterior stabilized rotating platform (PS RP).

Treatment assignment in this study is not randomized. Each site will only enroll patients in one of the four knee configuration sub-groups most commonly used as their standard of care.

This study allowed for enrolment into the study by two methods. The first method was by enroling subjects to receive the implant under study with the expectation to follow them out to 15 years. The second method was done to offset follow-up attrition. The second method allowed additional interested sites that had previously participated in a two-year follow-up study (NCT01746524) on this implant (subjects implanted and followed for two years) to reconsent interested subjects to be further followed out to 15 years in this study. The original 29 sites enroled 1232 subjects. Adding of the interested sites from the 2-yr follow-up study (NCT01746524) increased the sites from 29 to 37 sites. As of the last study update, the current enrolment is now1538.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female and between the ages of 22 and 75 years at the time of surgery, inclusive.
* Subject was diagnosed with NIDJD.
* Subject is a suitable candidate for cemented primary total knee arthroplasty using the devices described in this protocol with either resurfaced or non-resurfaced patellae.
* Subject has given voluntary, written informed consent to participate in this clinical investigation and has authorized the transfer of his/her information to DePuy.
* Subject is currently not bedridden.
* Subject in the opinion of the Clinical Investigator, is able to understand this clinical investigation and is willing and able to perform all study procedure and follow-up visits and co-operate with investigational procedures.
* Subject must be comfortable with speaking, reading and understanding questions and providing responses in an available translated language for the PROs in the protocol.
* The devices specified in this protocol were implanted.

Exclusion Criteria:

* Subject is a woman who is pregnant or lactating.
* Contralateral knee has already been enrolled in this study.
* Subject had a contralateral amputation.
* Previous partial knee replacement (unilateral, bicompartmental or patellofemoral joint replacement), patellectomy, high tibial osteotomy or primary TKA in affected knee.
* Subject is currently experiencing radicular pain from the spine.
* Subject has participated in an IDE/IND clinical investigation with an investigational product in the last three months.
* Subject is currently involved in any personal injury litigation, medical-legal or worker's compensation claims.
* Subject is a known drug or alcohol abuser or has a psychological disorder that could affect their ability to complete patient reported questionnaires.
* Subject was diagnosed with fibromyalgia that is currently being treated with prescription medication.
* Subject has significant neurological or musculoskeletal disorders or disease that may adversely affect gait or weight bearing (e.g. muscular dystrophy, multiple sclerosis, Charcot disease).
* Subject is suffering from inflammatory arthritis (e.g. rheumatoid arthritis, juvenile rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosis, etc.).
* Subject is not comfortable with speaking, reading, and understanding questions and providing responses in an available translated language for the PROs in the protocol.
* Subject has a medical condition with less than 5 years of life expectancy.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1542 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2030-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Survivorship of each configuration. | Minimum 15 years (5414 - 5658 days)
  Kaplan-Meier survival analysis will be used to calculate the survivorship of all 4 configurations (CR FB, CR RP, PS FB, PS RP).

SECONDARY OUTCOMES:
Survivorship | Minimum 5 years (1764 - 3588 days)
  Kaplan-Meier survival analysis will be used to calculate the survivorship of all 4 configurations (CR FB, CR RP, PS FB, PS RP).
Survivorship | Minimum 10 years (3589 - 5413 days)
  Kaplan-Meier survival analysis will be used to calculate the survivorship of all 4 configurations (CR FB, CR RP, PS FB, PS RP).
Implant fixation: Radiographic assessment of bone-implant interface performance | Minimum 1 year (304 - 668 days)
  Radiographic success is defined as: absence of progressive radiolucent lines greater than or equal to 2mm in any one zone; absence of lytic lesions in any zone; absence of individual component position change >3degrees in any plane.
Implant fixation: Radiographic assessment of bone-implant interface performance | Minimum 2 years (669 - 1763 days)
  Radiographic success is defined as: absence of progressive radiolucent lines greater than or equal to 2mm in any one zone; absence of lytic lesions in any zone; absence of individual component position change >3degrees in any plane.
Implant fixation: Radiographic assessment of bone-implant interface performance | Minimum 5 years (1764 - 3588 days)
  Radiographic success is defined as: absence of progressive radiolucent lines greater than or equal to 2mm in any one zone; absence of lytic lesions in any zone; absence of individual component position change >3degrees in any plane.
Implant fixation: Radiographic assessment of bone-implant interface performance | Minimum 10 years (3589 - 5413 days)
  Radiographic success is defined as: absence of progressive radiolucent lines greater than or equal to 2mm in any one zone; absence of lytic lesions in any zone; absence of individual component position change >3degrees in any plane.
Implant fixation: Radiographic assessment of bone-implant interface performance | Minimum 15 years (5414 - 5658 days)
  Radiographic success is defined as: absence of progressive radiolucent lines greater than or equal to 2mm in any one zone; absence of lytic lesions in any zone; absence of individual component position change >3degrees in any plane.
Patient Reported Outcome: EuroQol 5D 3L questionnaire (EQ-5D-3L) | Pre-op (-90 to -1 days before surgery), <1 year (1 - 303 days), minimum 1 year (304 - 668 days), minimum 2 years (669 - 1763 days), minimum 5 years (1764 - 3588 days), minimum 10 years (3589 - 5413 days), minimum 15 years (5414 - 5658 days).
  EuroQol 5D 3L questionnaire is a standardized instrument for use as a measure of health outcome that is designed for completion by the subject.
Patient-reported Outcome: Oxford Knee Score | Pre-op (-90 to -1 days before surgery), <1 year (1 - 303 days), minimum 1 year (304 - 668 days), minimum 2 years (669 - 1763 days), minimum 5 years (1764 - 3588 days), minimum 10 years (3589 - 5413 days), minimum 15 years (5414 - 5658 days).
  The Oxford Knee Score (OKS) is a patient self-administered 12-item questionnaire with each question having a Likert-lie response option. Each item is scored from 0 to 4, and the items are summated, with lower total scores indicating poorer performance. The OKS measures pain and general activities of daily living.
Patient-reported Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) | Pre-op (-90 to -1 days before surgery), <1 year (1 - 303 days), minimum 1 year (304 - 668 days), minimum 2 years (669 - 1763 days), minimum 5 years (1764 - 3588 days), minimum 10 years (3589 - 5413 days), minimum 15 years (5414 - 5658 days).
  The Knee injury and Osteoarthritis Outcome Score (KOOS) is a patient self-administered questionnaire that consists of 42 questions and includes the WOMAC Osteoarthritis index. The KOOS consists of 5 subscales; pain, other symptoms, activities of daily living (ADL), sport and recreational function and knee related quality of life. Each question has 5 Likert- like response options. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Patient-reported Outcome: Pre-surgical/Post-surgical Patient's Knee Implant Performance (PKIP) | Pre-op (-90 to -1 days before surgery), <1 year (1 - 303 days), minimum 1 year (304 - 668 days), minimum 2 years (669 - 1763 days), minimum 5 years (1764 - 3588 days), minimum 10 years (3589 - 5413 days), minimum 15 years (5414 - 5658 days).
  The Pre Surgical and/or Post-surgical Patient's Knee Implant Performance (PKIP) questionnaire is a patient self-administered questionnaire that consists of 25 questions relating to the patient's awareness of their knee. Questions include the patient's self-confidence about the current status of their knee performance, stability, and overall satisfaction. Each question has a 5, 6 or 10 Likert- like response option.
Patient-reported Outcome: Knee Society Score | Pre-op (-90 to -1 days before surgery), <1 year (1 - 303 days), minimum 1 year (304 - 668 days), minimum 2 years (669 - 1763 days), minimum 5 years (1764 - 3588 days), minimum 10 years (3589 - 5413 days), minimum 15 years (5414 - 5658 days).
  The Knee Society Score is a self-administered questionnaire. The subject completes questions regarding: Symptoms (3 questions), Patient Satisfaction (5 questions), Patient Expectations (3 questions), Functional Activities (5 questions), Standard Activities (6 questions), Advanced Activities (5 questions), and Discretionary Knee Activities ( 4 questions). Likert responses are used, typically with five response options.
Evaluate the impact of surgeon learning curve on clinical and functional outcomes | <1 year (1 - 303 days), minimum 1 year (304 - 668 days), minimum 2 years (669 - 1763 days), minimum 5 years (1764 - 3588 days), minimum 10 years (3589 - 5413 days), minimum 15 years (5414 - 5658 days).
  A surgeon learning curve will be investigated by comparing learning curve cases (the pooled cohort of each surgeon's first 10 study Subjects) with all investigational Subjects. All primary and secondary outcomes will be compared across the learning curve and post-learning curve Subject cohorts.
Evaluate changes in femoral component and tibial component alignment | Pre-op (-90 to -1 days before surgery), <1 year (1 - 303 days), minimum 1 year (304 - 668 days), minimum 2 years (669 - 1763 days), minimum 5 years (1764 - 3588 days), minimum 10 years (3589 - 5413 days), minimum 15 years (5414 - 5658 days).
  Radiographs will be reviewed by an independent radiographic reviewer (IRR) in order to minimize bias of radiographic outcomes. Data from the IRR radiographic evaluations will be used to evaluate femoral and tibial component alignment over time.
Type and Frequency of Adverse Events (AEs) for all enrolled subjects | Pre-op (-90 to -1 days before surgery), <1 year (1 - 303 days), minimum 1 year (304 - 668 days), minimum 2 years (669 - 1763 days), minimum 5 years (1764 - 3588 days), minimum 10 years (3589 - 5413 days), minimum 15 years (5414 - 5658 days).
  All Serious AEs must be reported to Sponsor. All device-related or procedure-related adverse events must be reported to Sponsor.

CONTACTS AND LOCATIONS:
Overall Officials: Allyson Morris, Study Director — DePuy Synthes
Locations (28):
- United States (10):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Orthopaedic Specialty Institute, Orange, California
  - Florida Research Associates, LLC, DeLand, Florida
  - Center for Hip and Knee Surgery, Mooresville, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Washington University School of Medicine, St Louis, Missouri
  - Orthopedic One, Columbus, Ohio
  - OrthoNeuro, New Albany, Ohio
  - Penn State Hershey Bone & Joint Institute, Hershey, Pennsylvania
  - Texas Institute for Hip and Knee Surgery, LLC, Austin, Texas
- Canberra Hospital-Trauma & Orthopaedic Research Unit, Adelaide, South Australia, Australia
- Austria (2):
  - Univ.-Klinik für Orthopädie, Vienna, Lower Austria
  - Krankenhaus der Barmherzigen, Linz, Upper Austria
- Monica Camputs O.L.V. Middelares, Antwerp, Belgium
- University of Western Ontario-Department of Orthopaedic Surgery, London, Ontario, Canada
- Germany (2):
  - Orthopädische Klinik für die Universität Regensburg, Bad Abbach, Bavaria
  - UniversitatsKlinikum Heidelberg, Heidelberg
- Queen Mary Hospital, Hong Kong, Hong Kong
- University Malaya Medical Centre, Kuala Lumpur, Malaysia
- Ascot Hospital, Auckland, New Zealand
- Singapore General Hospital-Dept of Orthopaedic Surgery, Singapore, Singapore
- South Korea (2):
  - Seoul National University Boramae Hospital, Seoul, Dongjak-gu
  - Seoul National University Hospital, Seoul
- United Kingdom (5):
  - Queen Mary Hospital, Dunfermline, Fife
  - Robert Jones & Agnes Hunt Orthopaedic Hospital, Gobowen, Oswestry
  - New Royal Infirmary of Edinburgh, Edinburgh, Scotland
  - Princess Alexandria Hospital, Harlow
  - Clifton Park NHS Treatment Centre, York